CLINICAL TRIAL: NCT01812668
Title: Pilot Trial of Oral Cabozantinib/XL184 in Metastatic Castrate Resistant Prostate Cancer to Explore the Changes in Bone and Tumor Imaging Related Pathways
Brief Title: Cabozantinib-S-Malate in Treating Patients With Hormone-Resistant Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-185; NCI-2013-00399 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; clevudine; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cabozantinib-s-malate) (Experimental): Patients receive cabozantinib-s-malate PO daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cabozantinib-s-malate; Radiation: fluorine F 18 d-FMAU; Procedure: positron emission tomography; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cabozantinib-s-malate — Given PO
  Other Names: BMS-907351; Cometriq; XL184
Radiation: fluorine F 18 d-FMAU — Undergo 18F PET/FMAU PET scan
Procedure: positron emission tomography — Undergo 18F PET/FMAU PET scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies cabozantinib-s-malate in treating patients with hormone-resistant metastatic prostate cancer. Cabozantinib-s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the timing, pathophysiology, and magnitude of changes in tumor imaging and pharmacodynamic markers with XL184 (cabozantinib-s-malate) treatment in metastatic castrate resistant prostate cancer.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) achieved with XL184 in metastatic castrate resistant prostate cancer (CRPC) patients.

II. To evaluate the feasibility of the therapy, and the toxicities associated. III. To evaluate overall survival (OS) in metastatic CRPC patients post androgen deprivation therapy (ADT) treated with XL-184.

OUTLINE:

Patients receive cabozantinib-s-malate orally (PO) daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histologically confirmed prostate adenocarcinoma with radiologic evidence of metastases
* If patient are on anti-androgens, these should be discontinued, at least 4 weeks prior for flutamide and at least 6 weeks for bicalutamide or nilutamide
* At least 14 days should have elapsed from prior radiation therapy to bone metastases from prostate cancer
* The patient has received a maximum of one prior chemotherapy regimen for metastatic prostate cancer
* Patients must demonstrate disease progression on or after most recent systemic therapy, either by prostate-specific antigen (PSA), new bone metastases or by measurable disease criteria per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines
* Patients should have received either luteinizing hormone-releasing hormone (LHRH) analogue, or LHRH analogue and anti- androgen for metastatic prostate cancer
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Bisphosphonate therapy can be continued if started prior to protocol enrollment
* Patients must have blood pressure (BP) readings < 150/90 prior to enrollment
* Absolute neutrophil count (ANC) >= 1500/mm^3 without colony stimulating factor support
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Bilirubin =< 1.5 x the upper limit of normal (ULN); for subjects with known Gilbert's disease, bilirubin =< 3.0 mg/dL
* Serum albumin >= 2.8 g/dl
* Serum creatinine =< 1.5 x ULN or creatinine clearance (CrCl) >= 50 mL/min; for creatinine clearance estimation, the Cockcroft and Gault equation should be used
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN if no liver involvement, or =< 5 x ULN with liver involvement
* Lipase < 1.5 x the upper limit of normal (except for subjects with adenocarcinoma of the pancreas)
* Urine protein/creatinine ratio (UPCR) =< 1
* Serum phosphorus >= lower limit of normal (LLN)
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Patients participating in this trial must also be eligible and willing to sign consent for participation in [2'-18F]-1-(2'-deoxy-2'-fluoro-beta-D-arabinofuranosyl)thymine (FMAU) and 18F-flouride positron emission tomography (PET) scans done under separate protocols
* Sexually active subjects (men) must agree to use medically accepted barrier methods of contraception (eg, male condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used by the female partner; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control
* Projected life expectancy of at least 6 months
* No prior history of other malignancies in the last 3 years, except for squamous and basal cell skin cancer

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (eg, cytokines or antibodies) within 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment
* Prior treatment with cabozantinib
* The subject has received radiation therapy:

  * To the thoracic cavity or gastrointestinal tract within 3 months of the first dose of study treatment
  * To bone or brain metastasis within 14 days of the first dose of study treatment
  * To any other site(s) within 28 days of the first dose of study treatment
* The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment; patients receiving LHRH or gonadotropin-releasing hormone (GnRH) agonists to maintain castrate levels of testosterone or patients on bisphosphonate/denosumab, may be maintained on these agents
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* The subject has a primary brain tumor
* The subject has active brain metastases or epidural disease (Note: Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible; neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment; baseline brain scans are not required to confirm eligibility)
* The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test results at screening >= 1.3 x the laboratory ULN
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor xabans (Xa) inhibitors, or antiplatelet agents (eg, clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* The subject has experienced any of the following within 3 months before the first dose of study treatment:

  * Clinically-significant hematemesis or gastrointestinal bleeding
  * Hemoptysis of >= 0.5 teaspoon (2.5 ml) of red blood
  * Any other signs indicative of pulmonary hemorrhage
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor in contact with, invading or encasing major blood vessels
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained BP > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment (BP must be controlled at screening)
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following at the time of screening

      * Intra-abdominal tumor/metastases invading gastrointestinal (GI) mucosa
      * Active peptic ulcer disease
      * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
    * Any of the following within 6 months before the first dose of study treatment:

      * History of abdominal fistula
      * Gastrointestinal perforation
      * Bowel obstruction or gastric outlet obstruction
      * Intra-abdominal abscess. Note: Complete resolution of an intraabdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months ago
    * GI surgery (particularly when associated with delayed or incomplete healing) within 28 days; Note: Complete healing following abdominal surgery must be confirmed prior to initiating treatment with cabozantinib even if surgery occurred more that 28 days ago
  * Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea and esophagus
  * Other clinically significant disorders such as:

    * Active infection requiring systemic treatment
    * Serious non-healing wound/ulcer/bone fracture
    * History of organ transplant
    * Concurrent uncompensated hypothyroidism or thyroid dysfunction
    * History of major surgery within 4 weeks or minor surgical procedures within 1 week before randomization
* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 470 ms within 28 days before randomization
* The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* The subject has had evidence within 2 years of the start of study treatment of another malignancy, which required systemic treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2019-01-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka Vaishampayan, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cabozantinib-s-malate)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 69 [56 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in PET Standard Uptake Value SUV Levels Pre-treatment to Post-treatment.
Description: Change in PET standard uptake value SUV levels (each value measured in g/ml). (post-treatment - pre-treatment)/pre-treatment x 100 , therefore, measured in percentage change from baseline.
Time Frame: Baseline to 4 weeks
Measure: Median (Full Range); unit: percentage change from baseline
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 20
percentage change from baseline | -56 [-85 to -5]

2. Secondary Outcome: Time to Progression
Description: Summarized via the Kaplan-Meier (K-M) survivorship estimate.
Time Frame: From date of registration to date of first documented disease progression, or death from any cause, assessed up to 1 year
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 20
months | 4.1 [2.3 to 5.3]

3. Secondary Outcome: Number of Participants With Indicated Toxicities Grade 3 or Higher
Description: Type of toxicities graded per National Cancer Institute (NCI) CTCAE version 4.0 Summarized via their frequency distribution and point estimate of the proportion.
Time Frame: Up to 4 weeks post-treatment, about 2 years on average.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 20
Participants
  Parkinson like syndrome | 1
  UTI | 1
  anemia | 2
  decreased ALC | 2
  decreased platelet | 1
  dehydration | 1
  diarrhea | 1
  fatigue | 3
  foot blisters | 1
  hyperglycemia | 2
  hypertension | 11
  hypophosphatemia | 2
  increased AST | 1
  mandibular abscess | 1
  mucositis | 1
  pleurisy | 1
  pneumonia | 1
  urinary retention | 1
  weight loss | 2

4. Secondary Outcome: Number of Participants With Indicated Clinical Response Based on the RECIST Criteria 1.1
Description: Number of Participants with Indicated Clinical response based on the RECIST criteria 1.1 summarized via their frequency distribution.
Time Frame: Up to 1 year
Population: Patients with measurable disease
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 9
Participants | 6

5. Secondary Outcome: PSA Response Based on the RECIST Criteria 1.1
Description: Summarized via their frequency distribution, point estimate of the proportion, and the Wilson type 80% CI.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 20
Participants | 8

6. Secondary Outcome: PET Response Based on the RECIST Criteria 1.1
Description: Summarized via their frequency distribution, point estimate of the proportion, and the Wilson type 80% CI.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 20
Participants | 19

ADVERSE EVENTS:
Time Frame: All untoward events that occur after start of therapy through 30 days after the last dose of study treatment are to be recorded, about 12 months on average.
Arm/Group | Treatment (Cabozantinib-s-malate)
All-Cause Mortality (participants affected / at risk) | 18/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib-s-malate) (N=20)
hand foot syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
urinary infection (Renal and urinary disorders) | 1 (1)
elevated creatinine (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib-s-malate) (N=20)
anemia (Blood and lymphatic system disorders) | 3 (3)
decreased ALC (Blood and lymphatic system disorders) | 2 (2)
GERD (Gastrointestinal disorders) | 2 (2)
UTI (Renal and urinary disorders) | 2 (2)
anorexia (Psychiatric disorders) | 14 (14)
blisters (Skin and subcutaneous tissue disorders) | 2 (2)
bone pain (Musculoskeletal and connective tissue disorders) | 6 (6)
chills (Metabolism and nutrition disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 9 (9)
dizziness (General disorders) | 2 (2)
dry mouth (General disorders) | 5 (5)
dysgeusia (Gastrointestinal disorders) | 6 (6)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
edema (Blood and lymphatic system disorders) | 5 (5)
fatigue (General disorders) | 17 (17)
hand/foot (Musculoskeletal and connective tissue disorders) | 3 (3)
headache (Nervous system disorders) | 4 (4)
hoarseness (General disorders) | 5 (5)
hyperglycemia (Endocrine disorders) | 2 (2)
hypertension (Vascular disorders) | 12 (12)
hypophosphatemia (Blood and lymphatic system disorders) | 2 (2)
hypothyroidism (Endocrine disorders) | 5 (5)
increased ALT (Blood and lymphatic system disorders) | 2 (2)
increased AST (Blood and lymphatic system disorders) | 4 (4)
mucositis (Gastrointestinal disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 10 (10)
rash (Skin and subcutaneous tissue disorders) | 6 (6)
urinary frequency (Renal and urinary disorders) | 3 (3)
urinary retention (Renal and urinary disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 4 (4)
weakness (General disorders) | 3 (3)
weight loss (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT01812668/Prot_SAP_000.pdf